CLINICAL TRIAL: NCT03911557
Title: Phase 2 Investigation of MEDI4736 (Durvalumab) and Tremelimumab Combination in Somatically Hypermutated Recurrent Solid Tumors
Brief Title: Durvalumab and Tremelimumab Combination in Somatically Hypermutated Recurrent Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John L. Villano, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, John L. Villano, MD, PhD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18-MULTI-25-PMC
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid
Keywords: mutational burden; TMB; PD-1; CTLA-4; MEDI4736; durvalumab; tremelimumab; immune therapy; refractory
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with moderate to high tumor mutational burden (Experimental): Patients with recurrent or refractory disease in solid tumors naïve to anti-PD-1/PD-L1 or anti-CTLA-4 immunotherapy and have moderate to high tumor mutational burden (TMB)
  Interventions: Drug: Durvalumab and Tremelimumab

INTERVENTIONS:
Drug: Durvalumab and Tremelimumab — Durvalumab 1500mg + tremelimumab 75mg via IV infusion Q4W, starting on Week 1, for up to a maximum of 4 doses/cycles followed by durvalumab monotherapy 1500 mg via IV infusion Q4W, starting 4 weeks after the last infusion of the combination, for up to a maximum of 2 years of total therapy.

SUMMARY:
This study will examine whether patients with relapsed/refractory solid tumors harboring evidence of somatic hypermutation (intermediate versus high tumor mutational burden) will exhibit improvement in disease progression-free survival with dual Tremelimumab and Durvalumab treatment.

DETAILED DESCRIPTION:
This study is phase II basket trial to evaluate the benefit of immunotherapy (Durvalumab and Tremelimumab combination) in treatment of relapse/refractory solid tumor patients whose tumors express a high tumor mutational burden (TMB high >20 mutations/MB) or moderate tumor mutational burden (10-20 mutations/MB) as based on next generation sequencing (NGS). The primary endpoint of the study is the TTP (time-to-progression) ratio or growth modulation index (GMI) which is defined for individual patients as the ratio of their TTP on the current therapy to their TTP on the most recent previous therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory solid tumor patients not previously treated with anti-PD-1/PD-L1 or anti-CTLA-4 immunotherapy whose tumors expressed a high tumor mutational burden (TMB) (TMB high >20 mutations/MB) or moderate TMB (10-20 mutations/MB) as based on next generation sequencing (NGS)
2. Age >18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of at least 2 and life expectancy greater than 3 months
4. Accurate documentation of date of starting previous therapy and date of progression to establish TTP from most recent therapy
5. Patient must have normal organ and marrow function independent of transfusion for at least 7 days prior to screening and independent of growth factor support for at least 14 days prior to screening as defined below:
6. Absolute neutrophil count (ANC ≥1.5 (or 1.0) x (> 1500 per mm3)
7. Platelet count ≥100 (or 75) x 109/L (>75,000 per mm3)
8. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome, who will be allowed only in consultation with their physician.
9. AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
10. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
11. The effects of MEDI4736 and tremelimumab on the developing human fetus are unknown. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
12. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
13. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
14. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception from the time of screening and must agree to continue using such precaution for 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy. Non-sterilized male partners of female patient must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.
15. Non-sterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 180 days after receipt of the final dose of durvalumab + tremelimumab combination therapy or 90 days after receipt of the final dose of durvalumab monotherapy. Not engaging in sexual activity is an acceptable practice; however, occasional abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
17. Body weight >30 kg
18. Cohort specific eligibility requirements:
19. Ability to undergo a fresh tumor biopsy for the purpose of screening for this clinical trial (including able and willing to give valid written consent) or the ability to access an available archival tumor sample taken less than 6 months prior to study enrollment if a fresh tumor biopsy is not feasible with an acceptable clinical risk and no antecedent treatment has been done.
20. MSS tumor as documented by either: IHC testing that does not suggest loss of MLH-1, MSH-2, PMS2 or MSH6. OR PCR testing that does not suggest MSI

Exclusion Criteria:

1. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapeutic agent, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) 30 days prior to the first dose of study drug
2. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician
3. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of the IP (investigational product, in this study, specifically durvalumab + tremelimumab combination). Note: Local surgery of isolated lesions for palliative intent is acceptable
4. History of allogenic organ transplantation
5. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
6. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
7. History of another primary malignancy except for

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of the IP ( durvalumab + tremelimumab combination ) and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
8. History of leptomeningeal carcinomatosis
9. Patients with untreated brain metastases, spinal cord compression, or leptomeningeal carcinomatosis should be excluded from this clinical trial because of their poor prognosis, because of symptoms that may arise form inflammatory reactions, and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images, both of which are obtained after treatment to the brain metastases. These imaging scans should both be obtained at least four weeks apart and show no evidence of intracranial progression). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of <10mg/day of prednisone or its equivalent and anti-convulsants for at least 14 days prior to the start of treatment
10. History of active primary immunodeficiency
11. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA
12. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
13. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
14. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab + tremelimumab combination therapy
15. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
16. Prior exposure to immune mediated therapy with anti-PD-1/ anti-PDL1including durvalumab therapy combined with an CTLA-4 therapy including tremelimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Time-to-progression ratio (TTP) | 2 years (baseline to follow-up)
  The TTP (time-to-progression) ratio is defined for individual patients as the ratio of their TTP on the current therapy to their TTP on the most recent previous therapy

SECONDARY OUTCOMES:
Progression-free survival | 2 years (baseline to follow-up)
  time to progression or death as measured from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Villano, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No